CLINICAL TRIAL: NCT01635816
Title: A Clinical Trial in Healthy Infants to Assess Lot-to-lot Consistency of Japanese Encephalitis Live Attenuated SA 14-14-2 Vaccine Manufactured in a New Good Manufacturing Practices Facility and Non-inferiority With Respect to an Earlier Product.
Brief Title: Immunogenicity of SA 14-14-2 JE Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PR-11050
Record Dates: First submitted 2012-07-04; First posted 2012-07-10 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2012-07

CONDITIONS: Healthy Infants
Keywords: Immunogenicity; SA 14-14-2 JE vaccine; Bangladesh

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- JE Vaccine existing facilities (Active Comparator): will receive JE live attenuated SA 14-14-2 vaccine manufactured in the existing facility (250 infants).
  Interventions: Biological: JE Vaccine existing facility
- JE vaccine new plant lot 1 (Active Comparator): Will receive Lot 1 JE live attenuated SA 14-14-2 vaccine manufactured in the new GMP facility (250 infants).
  Interventions: Biological: JE vaccine new plant lot 1
- JE vaccine new plant lot 2 (Active Comparator): Will receive Lot 2 JE live attenuated SA 14-14-2 vaccine manufactured in the new GMP facility (250 infants).
  Interventions: Biological: JE vaccine new plant lot 2
- JE vaccine new plant lot 3 (Active Comparator): Will receive will receive Lot 3 JE live attenuated SA 14-14-2 vaccine manufactured in the new GMP facility (250 infants).
  Interventions: Biological: JE vaccine new plant lot 3

INTERVENTIONS:
Biological: JE Vaccine existing facility — Will receive JE live attenuated SA 14-14-2 vaccine manufactured in the existing facility (250 infants).
  Arms: JE Vaccine existing facilities
Biological: JE vaccine new plant lot 1 — Will receive Lot 1 JE live attenuated SA 14-14-2 vaccine manufactured in the new GMP facility (250 infants).
  Arms: JE vaccine new plant lot 1
Biological: JE vaccine new plant lot 2 — Will receive Lot 2 JE live attenuated SA 14-14-2 vaccine manufactured in the new GMP facility (250 infants).
  Arms: JE vaccine new plant lot 2
Biological: JE vaccine new plant lot 3 — Will receive will receive Lot 3 JE live attenuated SA 14-14-2 vaccine manufactured in the new GMP facility (250 infants).
  Arms: JE vaccine new plant lot 3

SUMMARY:
The proposed Japanese Encephalitis (JE)Vaccine study is a four-arm double-blind randomized controlled single center trial to evaluate, by examining post-vaccination seroprotection titers, the lot-to-lot consistency of three lots of JE live attenuated SA 14-14-2 vaccine manufactured in a new GMP facility, and to establish non-inferiority of the new vaccine in comparison to a single lot of the same vaccine manufactured in the existing facility. The study will enroll a total of 1,000 Bangladeshi infants aged 10 to 12 months. In addition to providing immunogenicity data, JEV05 will provide local safety data of JE live attenuated SA 14-14-2 vaccine among Bangladeshi children. This will be the first step to secure licensure for this life-saving vaccine in Bangladesh as well as provide data to support WHO prequalification of JE live attenuated SA 14-14-2 vaccine.

DETAILED DESCRIPTION:
Vaccination is the most effective intervention to prevent JE and its associated morbidity and mortality (http://www.who.int.nuvi/Je/en). JE live attenuated SA 14-14-2 vaccine has been used in Asia for more than two decades in over 400 million children. Chengdu Institute of Biological Products (CDIBP), a Chinese manufacturer, has been producing JE live attenuated SA 14-14-2 vaccine since 1988. It has been demonstrated to be both safe and immunogenic in several observational and case-control studies providing protection for at least 5 years following a single dose. JE live attenuated SA 14-14-2 vaccine is licensed for use in China, India, Nepal, South Korea, Sri Lanka, and Thailand. Countries that have introduced JE vaccine into their national immunization programs have experienced dramatic reductions in JE incidence, leading WHO to declare vaccination the preferred JE control strategy.4

In order for JE live attenuated SA 14-14-2 vaccine to be available for purchase through UNICEF and GAVI for broader international use, including in Bangladesh, JE live attenuated SA 14-14-2 vaccine needs to undergo WHO prequalification. With technical support from PATH, CDIBP has established a new GMP facility, Building 208 JE production unit, maintaining WHO standards. A GMP Certificate for the new facility was issued on 11/16/2011. This certificate provides market authorization to distribute the new vaccine in China. To achieve WHO prequalification, JE live attenuated SA 14-14-2 vaccine produced in this new GMP facility needs to be shown to be similarly safe and immunogenic to JE live attenuated SA 14-14-2 vaccine produced in the existing facility, the JE viral vaccine production plant, and needs to demonstrate lot-to-lot consistency.

The proposed JEV05 study is a four-arm double-blind randomized controlled single center trial testing the immunogenicity of four lots of JE live attenuated SA 14-14-2 vaccine - three lots manufactured in the new GMP facility and one lot from the existing facility - in a total of 1000 Bangladeshi infants aged 10 to 12 months. The study will be conducted in the Matlab Health and Demographic Surveillance System (HDSS) intervention area, a rural site where many vaccine trials have been conducted.

A 5 ml blood sample will be collected from each child before vaccination and at 28 days post-vaccination. The sera will be tested using a plaque reduction neutralization test (PRNT) with JE neutralizing antibody titers > 1:10 considered seroprotective. The JEV05 trial will provide immunogenicity data on the three vaccine lots produced in the new GMP facility compared to a vaccine lot produced in the prior existing plant. It will also provide local immunogenicity and safety data of JE live attenuated SA 14-14-2 vaccine among Bangladeshi children. This will be the first step to secure licensure for this life-saving vaccine in Bangladesh as well as provide data to support WHO prequalification of JE live attenuated SA 14-14-2 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Infant's parent(s) or legal guardian(s) willing to provide signed informed consent.
* Healthy infants aged 10 to 12 months at enrollment residing in Matlab HDSS intervention area who have completed all doses of EPI immunizations (BCG, DPT, HBV, Hib, OPV and measles) at least 4 weeks prior to enrollment.

Exclusion Criteria:

* Acute medical illness with or without fever within the last 72 hours or an axillary temperature (≥ 37.5°C ) at the time of vaccination.
* Use of antibiotics or antipyretics within the last 72 hours prior to enrollment.
* Severely or moderately malnourished infants (<-3 Z score).
* History of prematurity (< 36 weeks of pregnancy).
* Underlying medical condition such as failure to thrive, inborn errors of metabolism, bronchopulmonary dysplasia, or any major congenital abnormalities requiring surgery or chronic treatment.
* History of serious chronic disease (e.g., cardiac, renal, neurologic, metabolic, rheumatologic, hematologic, or bleeding disorder).
* Known or suspected impairment of immunologic function.
* History of documented or suspected encephalitis or meningitis.
* History of seizures, including history of febrile seizures, or any other neurologic disorder.
* History of JE infection.
* Prior receipt of a JE vaccine.
* Received measles vaccine within 4 weeks prior to, or scheduled to receive a vaccination during, the conduct of this trial.
* Prior or anticipated receipt of immune globulin or other blood products, or injected or oral corticosteroids or other immune modulator therapy within 6 weeks of administration of the study vaccine.
* Serious adverse reactions (e.g. urticaria, angioedema, shock, breathlessness following vaccination or any life threatening condition) with any previous EPI vaccine.
* Unable to attend the scheduled visits or comply with the study procedures.
* Enrolled in another clinical trial involving any therapy.
* Any condition that in the opinion of the investigator, would pose a health risk to the child, or interfere with the evaluation of the study objectives.

Ages: 10 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of different lots of vaccines | 8 months
  JE immunogenicity will be parameterized as the percentage of children with demonstrated seroprotection (defined as a serum antibody titer of ≥ 1:10 as measured by PRNT) at 28 days post-immunization with JE live attenuated SA 14-14-2 vaccine.

CONTACTS AND LOCATIONS:
Locations (1):
- Matlab, Chāndpur, Bangladesh

REFERENCES:
- [Derived] Zaman K, Naser AM, Power M, Yaich M, Zhang L, Ginsburg AS, Luby SP, Rahman M, Hills S, Bhardwaj M, Flores J. Lot-to-lot consistency of live attenuated SA 14-14-2 Japanese encephalitis vaccine manufactured in a good manufacturing practice facility and non-inferiority with respect to an earlier product. Vaccine. 2014 Oct 21;32(46):6061-6. doi: 10.1016/j.vaccine.2014.09.012. Epub 2014 Sep 18. PMID 25239483